CLINICAL TRIAL: NCT04566874
Title: SPIRA™-A 3D Printed Titanium Anterior Lumbar Interbody Fusion Device and HCT/p Demineralized Bone Matrix Versus Medtronic Divergent™-L/Perimeter™ PEEK Anterior Lumbar Interbody Fusion Device and Recombinant Bone Morphogenic Protein-2
Brief Title: SPIRA™-A 3D and HCT/p DBM vs. Medtronic Divergent™-L/Perimeter™ and Recombinant BMP-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Camber Spine Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPA-2018
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis; Scoliosis
Keywords: lumbar spinal fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis; Scoliosis

STUDY DESIGN:
Intervention Model Description: single blind randomized 1:1
Who Masked: Participant
Masking Description: subjects will be blinded prior to surgery. Following surgery, maintaining masking may not be feasible as subjects will have access to medical records and/or radiographs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Spira-A with HCT/p DBM (Other): Single level Spira-A 3D printed Titanium ALIF Device with HCT/p DBM
  Interventions: Device: ALIF
- Medtronic PEEK ALIF with Infuse (Active Comparator): Single level Medtronic Divergent-L/Perimeter PEEK ALIF Device with Recombinant Bone Morphogenic Protein-2 (Infuse)
  Interventions: Device: ALIF

INTERVENTIONS:
Device: ALIF — Anterior Lumbar Interbody Fusion

SUMMARY:
A prospective, randomized, controlled clinical evaluation utilizing the SPIRA™ ALIF 3-D printed titanium interbody device with DBM vs a Medtronic PEEK ALIF interbody device with BMP

DETAILED DESCRIPTION:
This is a single blinded randomized 1:1, controlled, prospective clinical study to evaluate fusion status and patient reported outcomes in circumferential lumbar fusion between L2-S1 at a single level with posterior screw fixation (Camber Spine Orthros System) and anterior surgery consisting of one of the treatment groups: subjects treated with the SPIRA™-A Interbody Device and HCTP/p DBM or subjects treated with Medtronic Divergent-L or Perimeter™ PEEK ALIF Interbody Device and rhBMP-2 (6mg per level).

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature adults
* completed 6 month non-operative or conservative therapy
* signed informed consent
* back pain with radicular symptoms as evidenced by leg pain
* Degenerative Disc Disease involving a single level between L2 and S1
* subject willing to participate in study and follow protocol
* subject willing to comply with Post-op management program

Exclusion Criteria:

* systemic infection such as AIDS, HIV or Active hepatitis
* autoimmune disease
* significant metabolic disease that might compromise bone growth
* history of malignancy
* previous surgery for primary tumor, trauma or infection
* subject requires 2 or more levels of fusion
* previous spinal instrumentation or previous interbody fusion at involved level
* spondylolisthesis of grade greater than/equal to 2

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion | 6 months
  AP/Lateral, Flexion, Extension and CT radiographs
Radiographic Fusion | 12 months
  AP/Lateral, Flexion, Extension and CT radiographs
Radiographic Fusion | 24 months
  AP/Lateral, Flexion, Extension and CT radiographs

SECONDARY OUTCOMES:
Oswestry Disability Index | up to and including 24 months
  Improvement in the ODI as measured by a minimum of a 15 point improvement
Back and Leg VAS | up to and including 24 months
  Improvement in the VAS as measured by a minimum of a 20 point improvement.
VR-12 Health Survey | up to and including 24 months
  Improvement in the VR-12 Health Survey as demonstrated by pre-op and post-op evaluation
PROMIS score | up to and including 24 months
  Change in the PROMIS score

CONTACTS AND LOCATIONS:
Overall Officials: David Kaye, MD, Principal Investigator — Rothman Orthopaedic Institute
Locations (2):
- United States (2):
  - Rothman Orthopaedic Institure, Philadelphia, Pennsylvania
  - Texas Back Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No
data to be share with investigators only.